CLINICAL TRIAL: NCT07254884
Title: Safety and Efficacy of 2910 nm Fiber Laser Resurfacing and Laser-Coring Treatment to Lift the Eyebrow, Submental Lax Tissue and Address Advanced Signs of Facial Aging
Brief Title: Safety and Efficacy of 2910 nm Fiber Laser Resurfacing and Laser-Coring
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FA Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC 28-2025
Record Dates: First submitted 2025-10-01; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Rhytids; Skin Laxity
Keywords: Eyebrow Lift; Submental Tissue Lift; Wrinkles; Rhytids
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laser Treatment Arm (Experimental): Enrolled subjects will receive a series of two with an optional third 2,910 nm Fiber Laser treatments using fractional ablative resurfacing modes, laser-coring and full ablation addressing the full face and upper neck
  Interventions: Device: 2,910 nm mid-infrared erbium-doped fluoride fiber glass laser (UltraClear, Acclaro Medical)

INTERVENTIONS:
Device: 2,910 nm mid-infrared erbium-doped fluoride fiber glass laser (UltraClear, Acclaro Medical) — Enrolled subjects will receive a series of two with an optional third 2,910 nm Fiber Laser treatments using fractional ablative resurfacing modes, laser-coring and full ablation addressing the full face and upper neck.

SUMMARY:
The primary objective of this clinical trial is to evaluate the safety and effectiveness of the 2,910 nm mid-infrared erbium-doped fluoride fiber glass laser (UltraClear, Acclaro Medical) for non-invasive dermatological aesthetic treatment of three facial regions: eyebrow lift (Region 1), submental tissue lift (Region 2), and improvement of rhytids and skin laxity in the cheeks, midface, and jawline (Region 3).

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I-VI
* Male or female
* Subjects must be between 45 and 85 years of age
* Subjects must have the ability to receive two and up to three full face and upper neck resurfacing laser treatments (pending PI discretion) with desire to lift facial lax skin, submental and/or to lift the eyebrow area and/or improve facial wrinkles appearance
* Subjects must read, understand, and sign the Informed Consent Form
* Subjects must be willing and able to comply with all follow-up visit requirements
* Subjects must agree to refrain from using cosmeceutical agents or topical agents during the study, except as directed by study investigator
* Subjects must be rated as (2) Moderate Sagging to (4) Very Severe Sagging based on the Merz Scale: Jawline at Rest
* Subject identified as an appropriate candidate for study treatment based on principal investigator's opinion
* Subjects of childbearing potential have been on an acceptable form of contraception for 30 days prior to enrollment and agree to continue using throughout the course of the study

Exclusion Criteria:

* Subjects must not have active localized or systemic infections
* Subjects must not have a compromised ability for wound healing, such as: malnutrition, steroid use, history of collagen vascular disease (e.g., lupus, scleroderma, history of keloid scar formation), atopic dermatitis or immunologic abnormalities such as vitiligo
* Subjects must not be current smoker or have significant history of smoking
* Subjects must not have had treatments with systemic steroids or systemic retinoids in the 4-months prior to enrollment
* Subjects must not have had treatments with 5FU, diclofenac, imiquimod or PDT within 1-month prior to enrollment
* Subjects must not have severe or cystic facial acne; currently taking Accutane or have taken Accutane within the last 1-month
* Subjects must not have a known allergy to lidocaine or epinephrine, topical or injectable products containing lidocaine or any numbing medications
* Subjects must not have had previous surgery and/or fat transfer in the treatment area within the last 6-months
* Subject must not have had injectable soft tissue fillers within the last 12 months in the treatment area
* Subject must not have had Poly-L-Lactic acid (PLLA) fillers within the last 2 years in the treatment area
* Subject must not have had permanent filler i.e., Polymethylmethacrylate (PMMA) in the treatment area
* Subjects must not have had neurotoxins within the last 4-months in the treatment area
* Subject must not have a personal history of any facial threads i.e., PDO (Polydioxanone), PLLA (Polylactic acid), PCL (Polycaprolactone) in the treatment area within the last 12-months
* Subject must not have had a pulse dye or vascular laser, non-ablative laser, microneedling or RF microneedling treatments in the treatment area within the last 3-months
* Subject must not have had an ultrasound treatment such as HIFU, monopolar RF energy-based devices, ablative laser treatments in the treatment area within the last 6-months
* Subjects must not have a personal history of malignant melanoma, keloid scars, generalized psoriasis or systemic diseases that would preclude the use of topical anesthesia
* Subject must not have active sunburn or excessively tanned skin
* Subjects must not be pregnant or planning to become pregnant, have given birth less than 3 months ago, and/or breastfeeding during the study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Objective measurement of maximal eyebrow lift according to quantitative 2D imaging. | Six months following final treatment
Blinded Photographic Review | Six months following final treatment
  Blinded independent photographic review correct identification of pre-post image sequence for eyebrow lift, submental lift and improvement of lax skin in the lower face and submentum.
○ Objective measurement of lax submental tissue lift according to quantitative 2D imaging. | Six months following final treatment

SECONDARY OUTCOMES:
Physician rating on the Global Aesthetic Improvement Scale (PGAIS) | Six months following final treatment
  Physician graded aesthetic improvement, scored from photographs. Scale 0 - 4 with 4 being the most improved and 0 being worse than the original condition.
  4 - Very much improved, optimal cosmetic result, very significant improvement 3 - Much improved, market improvement in appearance from the initial condition, but not completely optimal, marked 2 - Improved, obvious improvement in appearance from the initial condition, but a pretreatment is needed, moderate
  1 - No change, the appearance is essential the same as the original condition in appearance from he initial condition 0 - Worse, the appearance is worse than the original condition, no improvement
Subjects rating on the Subject Global Aesthetic Improvement Scale & Satisfaction Questionnaire (SGAIS) | Six months following final treatment
  Subjects rate their perceived improvement of the treatment area on a 5 point scale.
  4- Very Much Improved, optimal cosmetic result, very significant improvement 3 - Much Improved, marked improvement in appearance from he initial condition but not completely optimal, marked 2 - Improved, obvious improvement in appearance from the initial condition, but a re-treatment is needed, moderate
  1 - No change, the appearance is essentially the same as the original condition in appearance from the initial condition 0 - Worse, the appearance is worse than the original condition, no improvement

OTHER OUTCOMES:
Evaluation of the pain and discomfort after treatment as reported by the subject on a visual analog scale (VAS) | Periprocedural and 15 minutes post-procedure
  VAS is a 10 point scale, reported by the subject. Subjects will be asked to report on a scale of 0-10, the average level of discomfort experienced during treatment.
  0 - No Pain
  5 - Moderate Pain
  10 - Unbearable Pain

IPD SHARING:
Plan to Share IPD: No